CLINICAL TRIAL: NCT03386630
Title: The Effects of Sufentanil or Morphine Added to Hyperbaric Bupivacaine in Spinal Anaesthesia for Elective Caesarean Section
Brief Title: Effects of Analgesics in Cesarean Section Elective
Acronym: CES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPS-CES-2017-01
Record Dates: First submitted 2017-11-20; First posted 2017-12-29 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Anesthesia; Functional
MeSH Terms: interventions — Sufentanil; Morphine

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial, without masking techniques, is proposed in pregnant women who are to undergo elective caesarean section by subarachnoid anesthesia with hyperbaric bupivacaine associated with sufentanil or morphine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperbaric bupivacaine+Sufentanil (Experimental): To evaluate in spinal anesthesia for elective cesarean section what association of hyperbaric bupivacaine 0.5% (0.06 mg Cm-1 in height) plus opioid: sufentanil (5 mcg)
  Interventions: Drug: Hyperbaric bupivacaine+Sufentanil
- Hyperbaric bupivacaine+morphine (Experimental): To evaluate in spinal anesthesia for elective cesarean section what association of hyperbaric bupivacaine 0.5% (0.06 mg Cm-1 in height) plus opioid: morphine (0,01 mg)
  Interventions: Drug: Hyperbaric bupivacaine+Morphine

INTERVENTIONS:
Drug: Hyperbaric bupivacaine+Sufentanil — To evaluate in spinal anesthesia for elective cesarean section what association of hyperbaric bupivacaine 0.5% (0.06 mg Cm-1 in height) plus opioid: sufentanil (5 mcg)
  Other Names: Sufentanil
  Arms: Hyperbaric bupivacaine+Sufentanil
Drug: Hyperbaric bupivacaine+Morphine — To evaluate in spinal anesthesia for elective cesarean section what association of hyperbaric bupivacaine 0.5% (0.06 mg Cm-1 in height) plus opioid: morphine (0,01 mg)
  Other Names: Morphine
  Arms: Hyperbaric bupivacaine+morphine

SUMMARY:
Two approved treatments for spinal anesthesia will be compared in women undergoing cesarean section.

It is usual to perform cesarean sections using spinal anesthesia with a local anesthetic (bupivacaine) plus some opioid, such as sufentanil or morphine. Both have been shown to decrease postoperative pain, but we try to check if one brings more benefit than the other.

ELIGIBILITY:
Inclusion Criteria:

* Patients of at least 18 years.
* Patients at least 36 weeks gestation.
* Patients scheduled for non-urgent cesarean section.
* Patients classified in the physical state of the American Society of Anesthesiologists (ASA) as grade I-II, and without important fetal pathological conditions.
* Signature of informed consent that allows them to be part of the study.

Exclusion Criteria:

* Pregnant women who reject the spinal technique.
* Patients with contraindication to spinal anesthesia.
* Patients with ASA> II classification.
* Patients with multiple pregnancy.
* Patients with three or more previous cesareans,
* Patients with BMI greater than or equal to 40 kg / m2.
* Language barrier.
* Patients with pre-eclampsia.
* Patients with a history of chronic pain.
* Patients with a history of psychiatric or drug abuse.
* Patients with allergy to any of the drugs used in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study population will be pregnant women who will undergo elective cesarean section through Subarachnoid anesthesia.
Enrollment: 66 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-28 (Actual)

PRIMARY OUTCOMES:
To evaluate the time it takes the patients administer a first analgesic bolus of morphine intravenous personally after subarachnoid anesthesia in elective cesarean section. | 3 days
  To evaluate in spinal anesthesia for elective cesarean section what association of hyperbaric bupivacaine plus opioid: sufentanil or morphine, produces a longer time for the patient to administer a first analgesic bolus of intravenous morphine.

SECONDARY OUTCOMES:
Lower intravenous morphine consumption | 24 hours after surgery
Levels of minor pain verbal scales | At 3, 6, 12 and 24 hours after surgery
  The measure is based in EVA (Escala visual analógica del dolor) scale. EVA scale allows to measure the pain intensity that the patient describes with the maximum reproducibility among the observers.
  1. Mild pain if the patient scores the pain as less than 3.
  2. Moderate pain if the assessment is between 4 and 7.
  3. Severe pain if the assessment is equal to or greater than 8.
Beginning of sitting and standing | At 48 hours after surgery
Mother´s side effects with respect to hemodynamic alteration, nausea, vomits, pruritus, tremor, urinary retention, sedation, respiratory depression, headaches, motor deficits, permanent sensory or autonomic deficits. | At intraoperative

OTHER OUTCOMES:
Values in the Apgar test | At 1 and 5 minutes after birth

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital La Línea, Cadiz, Spain